CLINICAL TRIAL: NCT03399331
Title: "The Efficacy of Honey or Olive Oil on the Severity and Pain of Oral Mucositis Compared to Placebo (Standard Care) in Children With Leukemia Receiving Intensive Chemotherapy
Brief Title: Honey or Olive Oil for Treating Oral Mucositis in Children and Adults With Leukemia Receiving Intensive Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Azusa Pacific University (Other); Daisy Foundation (Other)
Responsible Party: Principal Investigator, Lina Kordahi, Professor, leader for Research, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUR.LB.08
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Oral Mucositis; Leukemia
Keywords: honey, olive oil, oral mucositis, pain
MeSH Terms: conditions — Stomatitis; Leukemia; Pain | interventions — Olive Oil; Control Groups

STUDY DESIGN:
Intervention Model Description: three groups randomized using a computer generted number sequence
Who Masked: Investigator, Outcomes Assessor
Masking Description: Pain scores of the oral mucosa will be conducted twice a daily for study purposes. The patients will be assessed by their RNs for pain which is documented in the patient charts twice per day in the morign and in the evening (even in the absence of pain), the nurses will have no knowlegde of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): Efficacy of Manuka honey on severity and pain of OM compared to placebo (standard care) and to assess which of the two interventions is more beneficial.
  Interventions: Dietary Supplement: Manuka honey
- Group 2 (Experimental): Efficacy of olive oil on severity and pain of OM compared to placebo (standard care) and to assess which of the two interventions is more beneficial.
  Interventions: Dietary Supplement: olive oil
- Group 3 (Placebo Comparator): The control group at our institution is 5cc sodium bicarbonate, 5cc rinsidin and 5cc of mycostatin 4 times daily for children. For adults it is Caphosol in the BMT unit and in the Basile inpatient unit it is the magic solution (without xylocaine
  Interventions: Combination Product: Control group

INTERVENTIONS:
Dietary Supplement: Manuka honey — 5 for children or 10cc of honey for adults was ordered directly from a New Zealand company
  Arms: group 1
Dietary Supplement: olive oil — 5 cc of extra virgin olive oil for adults and 2 cc for children directly from a local distributor in south Lebanon will be given.
  Arms: Group 2
Combination Product: Control group — Control at our institution is 5cc sodium bicarbonate, 5cc rinsidin and 5cc of mycostatin 4 times daily for children. For adults it is Caphosol in the BMT unit and in the Basile inpatient unit it is the magic solution (without xylocaine).
  Arms: Group 3

SUMMARY:
Background: Oral mucositis (OM) is a significant complication occurring in approximately 40% of patients on chemotherapy regimens. Ulcerative lesions of OM can be very painful, with negative impact on diet, oral hygiene, and quality of life. Although a wide variety of agents have been tested to prevent OM or reduce its severity, none have provided conclusive evidence.

Objectives of this study will be: to determine the efficacy of honey or olive oil on the severity and pain of OM compared to placebo (standard care) and, (2) to assess which of the two interventions is more beneficial.

Research Questions:

1. Children/adults who receive honey (group 1) or olive oil (group 2) will have less severe OM compared to the control group (Severity is measured by recovery time from OM and is the primary outcome)
2. Children/adults who receive honey (group 1) OR Olive oil (group 2) will have less pain than the control group. (Severity of pain is the secondary outcome Methods: A randomized controlled study (RCT) will be used to evaluate the effect of topical application of honey or olive oil, in the treatment of chemotherapy-related OM in 60 participants with OM. The primary outcome will be the severity of mucositis, assessed by four trained nurses blinded to the study group using the scale presented by the World Health Organization (WHO). The secondary outcome will be pain also assessed by the four trained nurses on the visual analogue scale ort eh Wong Faces scale.

The relevance of this study lies in the possibility of challenging nurses in regard to the problem of OM and in proving a possible herbal cure that may influence clinical practice.

Data analysis: The characteristics of the three groups will be described using mean and SD, frequencies and percentages. Baseline differences between the two groups will be tested using ANOVA for continuous data, and the Chi-square for categorical data. Kruskall-Wallis (chi square) test will be used to find the association group assignment and WHO grades of OM and ANOVA and RANOVA tests will be used to find the association between group assignment and the pain scores. Bonferroni tests will be conducted to explore which of the three groups has the better outcomes.

DETAILED DESCRIPTION:
When parents or adults express interest in the study they will be approached by the Principal investigator (LKB) or the 2 research nurses (RS or RA) who will make contact with the children and their parents and explain the study, ,answer all their questions and concerns and inform them about the study benefits/potential risks (see recruitment script appendix B in proposal). If a parent approves to participate in the study, he/she will sign an informed consent and any child above 7 will be asked to sign an assent form. The investigator will also assure the parents that participation is totally voluntary and it is not a part of the conventional treatment and that they have the full right to refuse participating and withdraw from the study at any time, even after signing the consent.

Recruitment activities will take when the children are hospitalized at the Children's cancer center in Lebanon (CCCL), 8 North and the Bone Marrow unit (BMT). Patients, parents and children will also have access to flyers in the unit briefly explaining the study. Potential subjects will be identified through reviewing daily census on the inpatient unit of CCCL, 8 north or the BMT unit. Participates will be screened for eligibility and will be excluded if they have any condition that may affect the efficacy of treatment as listed in the exclusion criteria. Participants will be randomly assigned to 1 of 3 groups, 20 patients in each group. The randomization method will be prepared in advance by a statistician not involved in the study, using a paper list-generated random assignment sequencel. Based on group assignment, participants will receive a different compound applied topically to the oral mucosa 3 times daily until healing, or for 7 days, whichever comes first.

Group 1 will receive 10cc of honey for adults and 5 cc for children, which will be supplied directly from a New Zealand.

Group 2 will receive maximum 5 g of extra virgin olive oil for adults and 2 cc for children directly from a local distributor in south Lebanon. It will be stored in dark containers at room temperature for use in the study.

Group 3 will serve as control, which at our institution is 5cc sodium bicarbonate, 5cc rinsidin and 5cc of mycostatin 4 times daily for children. For adults it is Caphosol in the BMT unit and in the Basile inpatient unit it is the magic solution (without xylocaine).

Groups 1 and 2 patients will be instructed to slowly rinse the honey or olive oil in their mouths, swish it around for 1 minute duration, so as to make the honey or oil in contact with the oral mucosa and slowly swallow so as to make better contact with the pharyngeal mucosa. For group 3, patients will swish the respective solution for 1 minute then spit it out. The order of the different solutions will be written in each medical record by the attending physician and the nurse will observe the patient taking the solution and will document the administration on the hospital flowsheet.

The independent variable for this study is either olive oil or honey The dependent variables will be primary and secondary:

1. The primary outcome will be the severity of OM measured by recovery time, defined as the number of days from the initiation of treatment until healing or day 7 assessed by four trained nurses on a daily basis and who are blinded to the study group using the scale presented by the World Health Organization (WHO). The WHO scale is based upon the ability to eat and drink combined with objective signs of mucositis, namely erythema and ulceration (7). Visualisation of the oral cavity is critical for scoring, as the presence of oral ulcers delineates a WHO mucositis grade which ranges from 0 to 4 where higher scores correspond to worse mucositis. The WHO scale is classified as follows: grade 0=normal, no mucositis; grade 1=soreness and erythema; grade 2=erythema, ulcer, can eat solids; grade 3=ulcers, require liquid diet only; grade 4=alimentation not possible. The PI will establish inte-rater reliability with the four nurses by assessing patients on the WHO scale. Each nurse will conduct the assessment and compare her/his results with the PI, this will be done until a reliability of >. 80 is achieved. Reliability will be done before the study begins and then every month until the completion of the study.
2. The secondary outcome will be a pain assessed as per the institution's policy using the Visual analogue 10cm scale (VAS) or the Wong faces scale. A 0 indicates no mouth or throat pain and 10 indicates the most severe mouth or throat pain ( see appendix E in the proposal). The construct, convergent and predictive validity of the VAS and the Faces scales have been widely published (26). Pain scores of the oral mucosa will be conducted twice a daily for study purposes. The patients will be assessed by their RNs for pain which is documented in the patient charts twice per day in the morign and in the evening (even in the absence of pain).

ELIGIBILITY:
Inclusion Criteria:

The following are the inclusion criteria:

1. Children/Adults with leukemia (ALL, AML) receiving intensive (high dose) chemotherapy treatment such as myeloablative, doxorubicin or methotrexate during induction, consolidation and re-induction therapy.
2. Absence of any home remedy for mucositis
3. Patients with grades 1-3 OM based on the WHO grading system.

Exclusion Criteria:

1. Patients under non- intensive chemotherapeutic treatment.
2. Presence of advanced or severe periodontitis (patients with periodontal pockets of 6mm or more).
3. Patients with a cognitive disability which my no enable them to assess their pain
4. History of allergy to honey or olive oil.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The severity of Oral mucositis | 7 days or until healing or Discharge
  Defined as the number of days from the initiation of treatment until healing or day 7 assessed by four trained nurses on a daily basis and who are blinded to the study group using the World Health Organization (WHO) scale. The WHO scale is based upon the ability to eat and drink combined with objective signs of mucositis, namely erythema and ulceration. Visualisation of the oral cavity is critical for scoring, as the presence of oral ulcers delineates a WHO mucositis grade which ranges from 0 to 4 where higher scores correspond to worse mucositis. The PI will establish inte-rater reliability with the four nurses by assessing patients on the WHO scale. Each nurse will conduct the assessment and compare her/his results with the PI, this will be done until a reliability of >. 80 is achieved. Reliability will be done before the study begins and then every month until the completion of the study.

SECONDARY OUTCOMES:
Pain as reported by children | 7 days or until healing or Discharge
  Pain assessed as per the institution's policy using the Visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- American Univeristy of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
yes

REFERENCES:
- [Background] Al Jaouni SK, Al Muhayawi MS, Hussein A, Elfiki I, Al-Raddadi R, Al Muhayawi SM, Almasaudi S, Kamal MA, Harakeh S. Effects of Honey on Oral Mucositis among Pediatric Cancer Patients Undergoing Chemo/Radiotherapy Treatment at King Abdulaziz University Hospital in Jeddah, Kingdom of Saudi Arabia. Evid Based Complement Alternat Med. 2017;2017:5861024. doi: 10.1155/2017/5861024. Epub 2017 Feb 7. PMID 28270852
- [Background] Kobya Bulut H, Guducu Tufekci F. Honey prevents oral mocositis in children undergoing chemotherapy: A quasi-experimental study with a control group. Complement Ther Med. 2016 Dec;29:132-140. doi: 10.1016/j.ctim.2016.09.018. Epub 2016 Sep 19. PMID 27912937
- [Background] Xu JL, Xia R, Sun ZH, Sun L, Min X, Liu C, Zhang H, Zhu YM. Effects of honey use on the management of radio/chemotherapy-induced mucositis: a meta-analysis of randomized controlled trials. Int J Oral Maxillofac Surg. 2016 Dec;45(12):1618-1625. doi: 10.1016/j.ijom.2016.04.023. Epub 2016 Sep 3. PMID 27600797
- [Background] Jayalekshmi JL, Lakshmi R, Mukerji A. Honey on oral mucositis: A Randomized controlled trial. Gulf J Oncolog. 2016 Jan;1(20):30-7. PMID 27050177
- [Background] Cho HK, Jeong YM, Lee HS, Lee YJ, Hwang SH. Effects of honey on oral mucositis in patients with head and neck cancer: A meta-analysis. Laryngoscope. 2015 Sep;125(9):2085-92. doi: 10.1002/lary.25233. Epub 2015 Mar 16. PMID 25778825
- [Background] Hawley P, Hovan A, McGahan CE, Saunders D. A randomized placebo-controlled trial of manuka honey for radiation-induced oral mucositis. Support Care Cancer. 2014 Mar;22(3):751-61. doi: 10.1007/s00520-013-2031-0. Epub 2013 Nov 13. PMID 24221577
- [Background] Abdulrhman M, Elbarbary NS, Ahmed Amin D, Saeid Ebrahim R. Honey and a mixture of honey, beeswax, and olive oil-propolis extract in treatment of chemotherapy-induced oral mucositis: a randomized controlled pilot study. Pediatr Hematol Oncol. 2012 Apr;29(3):285-92. doi: 10.3109/08880018.2012.669026. PMID 22475306
- [Background] Song JJ, Twumasi-Ankrah P, Salcido R. Systematic review and meta-analysis on the use of honey to protect from the effects of radiation-induced oral mucositis. Adv Skin Wound Care. 2012 Jan;25(1):23-8. doi: 10.1097/01.ASW.0000410687.14363.a3. PMID 22218067